CLINICAL TRIAL: NCT02690727
Title: An Open Label, Randomized, Single Dose, Cross Over Study to Evaluate Food Effects on Relative Bioavailability of RP6530 Administered in Fasting and Fed Conditions in Healthy Volunteers
Brief Title: To Evaluate the Food Effect on Relative Bioavailability of RP6530 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rhizen Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RP6530-1501; ISI-P5-416 (Other: Algorithme Pharma Inc.)
Record Dates: First submitted 2016-02-15; First posted 2016-02-24 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2016-02

CONDITIONS: Healthy
Keywords: Fasting; Fed condition; Pharmacokinetics
MeSH Terms: conditions — Fasting | interventions — tenalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RP6530 in fast condition (Experimental): A single dose of RP6530 following fast condition
  Interventions: Drug: RP6530
- RP6530 in fed condition (Experimental): A single dose of RP6530 following fed condition
  Interventions: Drug: RP6530

INTERVENTIONS:
Drug: RP6530 — Single oral dose
  Other Names: A dual PI3K delta/gamma inhibitor

SUMMARY:
This is a single centre, open label, randomized, two-treatment, two-period, two-sequence, single dose crossover food effect study in 18 subjects. The subjects will receive the study medication under either fed or fast during each treatment period.

DETAILED DESCRIPTION:
The present study will be conducted in healthy male volunteers. A single oral dose will be administered to the subject in each treatment period (under either fasting or fed state). Each treatment period will be separated by at least 7 calendar days. Post dose PK blood samples will be collected in each treatment period to evaluate the food effect on bioavailability of RP6530. The safety and tolerability of single dose will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers; aged 18 to 45 years;
* Body mass index (BMI) between 18.0 and 30.0 kg/m2 inclusive, weight ≥ 50 kg;
* Non- smokers or ex-smokers;
* Able to give informed consent.

Exclusion Criteria:

* Subjects with evidence or history of clinically significant disease;
* Positive results to HIV Ag/Ab Combo, Hepatitis B surface Antigen (HBsAG (B) (hepatitis B)) or Hepatitis C Virus (HCV (C)) tests;
* Subjects who have received any investigational drug in the previous 28 days;
* Subjects participated in a study with PI3k inhibitors at least once in past year;
* Subjects who have received drugs metabolised by CYP3A4 enzyme in the previous 28 days.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, M.D, Principal Investigator — Algorithme Pharma Inc
Locations (1):
- Algorithme Pharma Inc, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- RP6530: Fast Condition First, Then Fed Condition: Fast Condition first, then Fed Condition
  RP6530: Single oral dose
- RP6530: Fed Condition First, Then Fast Condition: Fed Condition first, then Fast Condition
  RP6530: Single oral dose
Period: Overall Study
Arm/Group | RP6530: Fast Condition First, Then Fed Condition | RP6530: Fed Condition First, Then Fast Condition
Started | 9 | 9
Completed | 7 | 7
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 2

BASELINE CHARACTERISTICS:
Population: 18 healthy volunteers were enrolled to get at least 12 completed subjects to demonstrate food effect.
  * Safety population included all participants who received at least 1 dose of study drug.
  * PK population included all the participants who provided PK in both period.
Groups:
- All Participants: A single dose of RP6530 following fasting and Fed condition
  RP6530: Single oral dose
Arm/Group | All Participants
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 01
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Canada | 18
Weight [Mean (Standard Deviation); unit: Kg] | 73.9 (8.1)
Height [Mean (Standard Deviation); unit: cm] | 173.7 (7.2)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.50 (2.46)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Parameters (Area Under the Plasma Concentration Versus Time Curve (AUC))
Description: Pharmacokinetic parameters (Area under the plasma concentration versus time curve (AUC)) AUC0-T of RP6530 in fed and fast state.
Time Frame: up to 24 hours post-dose.
Population: subjects who provided evaluable data for both treatments (Fasting and fed conditions)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per millilitre (ng*h/mL)
Arm/Group | RP6530 in Fast Condition | RP6530 in Fed Condition
Number analyzed (Participants) | 14 | 14
nanogram*hour per millilitre (ng*h/mL) | 5277.01 (33.4) | 6726.99 (29.4)
Statistical Analysis 1: Comparison: RP6530 in Fast Condition vs RP6530 in Fed Condition; Test type: Superiority or Other; p = 0.0002, ANOVA; Ratio (%) = 128.49, 90% CI 2-sided [119.13 to 138.59]

2. Secondary Outcome: Number of Participants Who Were Evaluated for Adverse Events
Description: Number of Participants Who Were Evaluated for Adverse Events as Assessed by CTCAE v4.0
Time Frame: 7 days
Population: Healthy volunteers
Measure: Count of Participants; unit: Participants
Arm/Group | RP6530 in Fast Condition | RP6530 in Fed Condition
Number analyzed (Participants) | 16 | 16
Participants | 16 | 16

3. Secondary Outcome: Pharmacokinetic Parameters
Description: Peak Plasma Concentration (Cmax)
Time Frame: up to 24 hours post-dose.
Population: Subjects who provided evaluable data for both treatments
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per millilitre (ng/mL)
Arm/Group | RP6530 in Fast Condition | RP6530 in Fed Condition
Number analyzed (Participants) | 14 | 14
nanogram per millilitre (ng/mL) | 1311.77 (42.0) | 1753.78 (32.6)
Statistical Analysis 1: Comparison: RP6530 in Fast Condition vs RP6530 in Fed Condition; Test type: Superiority or Other; p = 0.0278, ANOVA; Ratio (%) = 139.27, 90% CI 2-sided [111.01 to 174.73]

ADVERSE EVENTS:
Time Frame: Day 1 to Day 7
Description: Subjects who entered the study and received at lease one of the treatments under study.
  2 HV dropped in 2nd period in "Fast Condition first, then Fed Condition sequence" similarly, two HV dropped in second period in "Fed Condition first sequence", therefore each treatment had 16 HV for AE evaluation; Fasting 16 and fed 16
Arm/Group | RP6530 in Fast Condition | RP6530 in Fed Condition
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 5/16 | 5/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RP6530 in Fast Condition (N=16) | RP6530 in Fed Condition (N=16)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Vessel puncture site bleeding (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
vessel puncture site swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 2 (2)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other